CLINICAL TRIAL: NCT03147014
Title: Cardiovascular Response to Maternal Hyperoxygenation in Fetal Congenital Heart Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, He Yihua,MD, Director of Department of Ultrosound, Beijing Anzhen Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MH-FCHD01
Record Dates: First submitted 2017-05-04; First posted 2017-05-10 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Hypoplastic Left Heart Syndrome; Aortic Coarctation; Atrial Septal Aneurysm
Keywords: Echocardiography; Congenital Heart Disease; Maternal hyperoxygenation
MeSH Terms: conditions — Hypoplastic Left Heart Syndrome; Aortic Coarctation; Heart Defects, Congenital

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Maternal Hyperoxygenation (Other): Maternal hyperoxygenation will be offered by administering 10 liters nasal cannula by face-mask (approximately 60% fiO2) for a minimum of 10 minutes.
  Interventions: Biological: Maternal hyperoxygenation

INTERVENTIONS:
Biological: Maternal hyperoxygenation — approximately 10-15 minutes of maternal hyperoxygenation

SUMMARY:
Cardiovascular Response to Maternal Hyperoxygenation in Fetal Congenital Heart Disease

DETAILED DESCRIPTION:
The purpose of this study is to investigate the phenomenon of cardiovascular system response to maternal hyperoxygenation in the fetus with congenital heart disease(CHD), which can provide further insight into fetal adaptations to CHD and improve our understanding of the pathophysiology of these conditions.Cases are gravidas with fetal congenital heart disease diagnosed by echocardiography various gestational weeks.The baseline fetal echocardiography parameters has obtained from these gravidas.Then the participants received 10-15 minutes hyperoxygenation, and the accordingly fetal echocardiography parameters were obtained.The objective of the study includes:(1)To investigate the response of the MCA PI to maternal hyperoxygenation in various forms of CHD. Middle cerebral artery(MCA) pulsatility index (PI) at MH will be compared to baseline at various gestational ages in a variety of types of CHD;(2)To investigate the response of the umbilical artery (UA) PI to maternal hyperoxygenation in various forms of CHD. UA PI at MH will be compared to baseline at various gestational ages in a variety of CHD; (3)To study the response of myocardial diastolic function to MH in various forms of CHD. Diastolic inflow patterns across the tricuspid and mitral valves will be measured and ductus venosus flow pattern will be evaluated at MH and compared to baseline at various gestational ages in a variety of CHD;(4)To investigate for any changes in cardiac output and the ratio of flow between the right and left ventricles in response to MH in various forms of CHD;(5)To investigate for changes in flow pattern at the aortic isthmus in those with suspicion or clear evidence of coarctation of the aorta.

ELIGIBILITY:
Inclusion Criteria:

* All singleton fetuses with CHD at all gestational ages are eligible for enrollment in the study. Patients will be recruited to enroll in the study as they present for clinical care at Fetal Echocardiography clinic. MH assessments will all be performed only at the Beijing Anzhen Hospital. Baseline room air data for CHD may be collected from other referring centers within the Anzhen network.

Exclusion Criteria:

* Non-sinus rhythm, presence of arrhythmia; Fetal hydrops; Severe brain anomaly (which may influence MCA flow); Evidence for significant ventricular dysfunction; Evidence for constriction of the ductus arteriosus

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
MCA PI change before and after maternal hyperoxygenation | 10-15 minutes
  The response of the MCA PI to maternal hyperoxygenation in various forms of CHD. MCA PI at MH will be compared to baseline at various gestational ages in a variety of types of CHD.

SECONDARY OUTCOMES:
UA PI change before and after maternal hyperoxygenation | 10-15 minutes
  Response of the umbilical artery (UA) PI to maternal hyperoxygenation in various forms of CHD. UA PI at MH will be compared to baseline at various gestational ages in a variety of CHD.

OTHER OUTCOMES:
Response of myocardial diastolic function to MH in various forms of CHD | 10-15 minutes
  Diastolic inflow patterns across the tricuspid and mitral valves will be measured and ductus venosus flow pattern will be evaluated at MH and compared to baseline at various gestational ages in a variety of CHD.
Systolic function change before and after MH | 10-15 minutes
  any changes in cardiac output and the ratio of flow between the right and left ventricles in response to MH in various forms of CHD.
Changes in flow pattern at the aortic isthmus | 10-15 minutes
  Changes in flow pattern at the aortic isthmus in those with suspicion or clear evidence of coarctation of the aorta

CONTACTS AND LOCATIONS:
Overall Officials: Yihua He, MD, Study Director — Beijing Anzhen Hospital
Locations (1):
- Beijng Anzhen Hospital, Beijing, Beijing Municipality, China